CLINICAL TRIAL: NCT00323609
Title: A Multicenter, Randomized, Prospective Clinical Trial to Compare the Short- and Long-term Safety and Effectiveness of Balloon Kyphoplasty to Vertebroplasty in the Treatment of Painful, Acute Osteoporosis-related Vertebral Body Compression Fractures (VCFs).
Brief Title: KAVIAR Study - Kyphoplasty And Vertebroplasty In the Augmentation and Restoration of Vertebral Body Compression Fractures
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to high number of patients terminating study early, low patient enrollment and difficulty in patient/investigator willingness for randomization
Sponsor: Medtronic Spine LLC (Industry)
Responsible Party: Sponsor
Organization: Medtronic Spinal and Biologics (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SP0601-KAVIAR
Record Dates: First submitted 2006-05-05; First posted 2006-05-09 (Estimated); Results first posted 2012-08-08 (Estimated); Last update posted 2018-01-02 (Actual); Status verified 2012-06

CONDITIONS: Vertebral Body Compression Fractures
Keywords: Kyphoplasty; Vertebroplasty; Balloon Kyphoplasty; Inflatable Bone Tamp; Spine; Back Pain; Vertebral Compression Fracture; Vertebral Body Compression Fracture
MeSH Terms: conditions — Back Pain | interventions — Vertebroplasty; Kyphoplasty

ARMS (2):
- Kyphoplasty (Active Comparator)
  Interventions: Procedure: Kyphoplasty
- Vertebroplasty (Active Comparator)
  Interventions: Procedure: Vertebroplasty

INTERVENTIONS:
Procedure: Vertebroplasty — Vertebroplasty involves placement of a needle into the vertebral body. Cement is injected into the vertebral body.
  Arms: Vertebroplasty
Procedure: Kyphoplasty — Balloon Kyphoplasty involves two inflatable bone tamps placed into the vertebral body in the spine. After the tamps are removed, the void is filled with viscous bone cement.
  Arms: Kyphoplasty

SUMMARY:
Patients with osteoporotic vertebral body compression fractures will be randomly assigned to treatment with balloon kyphoplasty or vertebroplasty. Over 2 years of follow-up, back pain, back function, quality of life, adverse events, subsequent fractures and cumulative healthcare costs will be compared.

DETAILED DESCRIPTION:
Medtronic Spine LLC is sponsoring the KAVIAR study, a randomized clinical trial comparing balloon kyphoplasty to vertebroplasty for the treatment of osteoporotic vertebral body compression fractures (VCFs). Up to 1,234 subjects at up to 75 study centers with one to three VCFs and VB morphologies suitable for both balloon kyphoplasty and vertebroplasty will be randomly assigned to receive one or the other procedure. Study visits will occur at baseline, 30 days postoperatively, and at 3, 12 and 24 months postoperatively. At all visits, adverse events, back pain, back function and quality of life will be assessed. In addition, a 7-day phone call will be conducted, which will include assessment of back pain, narcotic use and adverse events. At baseline, pre-discharge, 3-, 12- and 24-month visits, lateral spine x-rays will be taken. The primary endpoint will be the proportion of patients with one or more subsequent fractures at 12 and 24 months, detected radiographically as determined by a core radiology laboratory. Secondary clinical endpoints include changes from baseline in back pain, back function and quality of life, and adverse events. Secondary radiographic comparisons include the restoration and maintenance of VB height and angulation, and sagittal vertical axis, a measure of global sagittal balance. A postoperative CT scan will be evaluated to detect cement extravasation and to examine the relationship between cement distribution and clinical outcomes. Another important feature of the study is a detailed healthcare utilization data assessment. Combined with a costing methodology based on Medicare cost data and other sources, cumulative two-year healthcare costs related to VCF will be estimated. Combined with quality of life measurements, the cost analysis will allow a calculation of the relative cost-effectiveness of balloon kyphoplasty and vertebroplasty. Sample size is based on the primary endpoint, the proportion with subsequent fractures at 12 and 24 months.

ELIGIBILITY:
Inclusion Criteria

All subjects must meet all of the following criteria to be enrolled into the study:

1. Age > 21
2. 1 to 3 target VCFs meeting the following criteria:

   1. Fracture due to diagnosed or presumed underlying primary or secondary osteoporosis
   2. All target VCFs are between T5 and L5
   3. All target VCFs to be treated show either: i. Height change: An acute (< 6 month) change in VB height or morphology from a previous x-ray, CT or MRI, with height loss at the anterior, middle or posterior portion of the VB consistent with a worsening of 1 or more grades by the Genant criteria (17), OR ii. Positive MRI or bone scan: VB shows hyperintense signal on STIR sequence MRI or target VB is positive on radionuclide bone scan
   4. All VCFs to be treated have fracture age (time from pain onset to evaluation by the Investigator) of 6 months or less
   5. Back pain correlating with the location of at least one VCF
3. Treatment of all target VCFs is technically feasible by and clinically appropriate for BOTH vertebroplasty and balloon kyphoplasty. (Team approach only: Both the vertebroplasty and balloon kyphoplasty physician have reviewed radiographic studies and agree to this prior to enrolling the subject in the study.)
4. Pre-treatment back pain by numerical rating scale (NRS) score > 4 (0-10 scale)
5. Pre-treatment Oswestry Disability Index >20 (0 - 100 scale)
6. Subject states availability for all study visits
7. Subject is able to understand the risks and benefits of participating in the study and is willing to provide written informed consent
8. Subject has mental capacity to comply with the protocol requirements for 2-year duration of study

Exclusion Criteria

Subjects who meet any of the following conditions may not be enrolled into the study:

1. VB morphology or configuration is such that either balloon kyphoplasty OR vertebroplasty is not technically feasible for the targeted VCFs
2. Fracture due to high-energy trauma
3. Suspected OR proven cancer inside index vertebral body. Note that patients with chemotherapy-related osteoporosis may be included.
4. Disabling back pain due to causes other than acute fracture (e.g., sacroiliac fracture, symptomatic degenerative disc disease, lumbar spinal stenosis)
5. Any painful VCF with fracture age > 6 months
6. Any objective evidence of neurologic compromise at baseline
7. Previous balloon kyphoplasty or vertebroplasty for any VCF
8. Spine stabilization beyond balloon kyphoplasty or vertebroplasty required for targeted VCFs
9. Significant clinical comorbidity that may potentially interfere with long-term data collection or follow-up (e.g., dementia, severe comorbid illness)
10. Pre-existing conditions contrary to either balloon kyphoplasty or vertebroplasty, such as:

    1. Irreversible coagulopathy or bleeding disorder. Note regarding reversible coagulopathies: Subjects on coumadin or other anticoagulants may participate. Investigators should follow routine practices for perioperative discontinuation and re-initiation of anticoagulants.
    2. Allergy to any device materials (e.g., bone cement) for balloon kyphoplasty or vertebroplasty. Note that in subjects with allergy to iodine-based contrast, other non-iodine contrast solutions may be used.
    3. Any evidence of VB or systemic infection
11. Pregnant or child-bearing potential

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 404 (Actual)
Dates: Start 2006-08; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Reginald Knight, MD, Principal Investigator — Orthopedics International
Locations (26):
- United States (25):
  - Scottsdale Medical Imaging, Ltd, Scottsdale, Arizona
  - Minimally Invasive Surgical Solutions, San Jose, California
  - Torrance Memorial Medical Center, Torrance, California
  - Western Slope Study Group, Grand Junction, Colorado
  - The Center for Spinal Disorders, Tampa, Florida
  - Radiology Associates of Atlanta, Atlanta, Georgia
  - Ochsner Medical Center, New Orleans, Louisiana
  - William Beaumont Hospital, Royal Oak, Michigan
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Northwest Research & Educational Institute, Billings, Montana
  - Renown Regional Medical Center, Reno, Nevada
  - University Orthopedics, Rochester, New York
  - Atrium Medical Center, Franklin, Ohio
  - The Toledo Hospital, Toledo, Ohio
  - Clinical Radiology of Oklahoma, Edmond, Oklahoma
  - The Center for Orthopedic and Neurosurgical Care and Research (The Center), Bend, Oregon
  - Reading Hospital, Reading, Pennsylvania
  - The Methodist Hospital Research Institute, Houston, Texas
  - Scott & White Memorial Hospital, Temple, Texas
  - Intermountain Medical Center, Murray, Utah
  - Utah Valley Regional Medical Center, Provo, Utah
  - Carilion Roanoke Memorial Hospital, Roanoke, Virginia
  - St. Mary's Hospital, Huntington, West Virginia
  - Aurora Burlington Memorial Hospital, Burlington, Wisconsin
  - Aurora St. Luke's Medical Center, Milwaukee, Wisconsin
- Royal Victoria Hospital, Barrie, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- Kyphoplasty: This group of patients has received balloon kyphoplasty procedure.
- Vertebroplasty: This group of patients has received vertebroplasty procedure.
- Kyphoplasty Not Treated Patients; Vertebroplasty Not Treated Patients: Patients who met the enrollment criteria at screening and were randomized to treatment group had terminated prior to surgery or those who no longer met the inclusion criteria prior to surgery.
Period: Overall Study
Arm/Group | Kyphoplasty | Vertebroplasty | Kyphoplasty Not Treated Patients | Vertebroplasty Not Treated Patients
Started | 191 | 190 | 8 | 15
Completed | 100 (Revision retains subjects with follow-up data in a visit window when terminated in same visit window) | 91 (Revision retains subjects with follow-up data in a visit window when terminated in same visit window) | 0 | 0
Not Completed | 91 | 99 | 8 | 15
Not completed — Death | 16 | 21 | 0 | 0
Not completed — Lost to Follow-up | 9 | 10 | 0 | 0
Not completed — Physician Decision | 2 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 11 | 23 | 4 | 4
Not completed — Other non-VCF-related medical condition | 3 | 2 | 0 | 0
Not completed — Sponsor discontinued trial | 29 | 29 | 0 | 0
Not completed — Unrelenting or severe back pain | 1 | 1 | 0 | 0
Not completed — Logistical withdrawal | 9 | 5 | 0 | 1
Not completed — Other reason | 11 | 8 | 4 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Kyphoplasty | Vertebroplasty | Total
Number analyzed (Participants) | 191 | 190 | 381
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.5 (10.3) | 75.7 (10.5) | 75.6 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 151 | 144 | 295
  Male | 40 | 46 | 86
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 2 | 3
  Black or African American | 3 | 4 | 7
  Hispanic | 8 | 2 | 10
  White | 178 | 181 | 359
  Other | 1 | 0 | 1
Current Weight [Mean (Standard Deviation); unit: lbs] | 154.0 (40.2) | 160.2 (42.9) | 157.1 (41.6)
Current Height [Mean (Standard Deviation); unit: inches] | 63.8 (4.3) | 64.5 (4.0) | 64.1 (4.2)
Smoking Habit [Number; unit: participants]
  Never Smoked | 92 | 84 | 176
  Former Smoker | 68 | 84 | 152
  Current Smoker | 31 | 22 | 53
Osteoporosis Cause [Number; unit: participants]
  Suspected or confirmed primary osteoporosis | 179 | 172 | 351
  Suspected or confirmed secondary osteoporosis | 12 | 18 | 30
Number of patients with intend to treat VCFs [Number; unit: participants]
  One level of VCFs intend to treat | 149 | 150 | 299
  Two levels of VCFs intend to treat | 33 | 32 | 65
  Three levels of VCFs intend to treat | 9 | 8 | 17

OUTCOME MEASURES:

1. Primary Outcome: Percent of Subjects With One or More Subsequent Radiographic Fractures at 12 Months
Time Frame: 12 months
Population: Intent to treat population comprised of all subjects randomized and had initial treatment carried out. The n for each group with available data at 12-months is indicated.
Measure: Number; unit: percentage of participants
Arm/Group | Kyphoplasty | Vertebroplasty
Number analyzed (Participants) | 140 | 131
percentage of participants
  No subsequent VCF | 64.3 | 56.5
  One or more subsequent VCFs | 35.7 | 43.5
Statistical Analysis 1: Comparison: Kyphoplasty vs Vertebroplasty; Test type: Superiority or Other; p = 0.214, Fisher Exact

2. Secondary Outcome: Back Pain
Description: Back pain was assessed on a 10-point Numerical Rating Scale (NRS) from 0 (no pain) to 10 (worst possible pain).
Time Frame: 7 days, 30 days, 3 months, 12 months, 24 months post-operation
Population: Intent to treat population comprised of all subjects randomized and had initial treatment carried out. The n for each group with available data at each time point are indicated; for subjects who have secondary surgery, the last value before the first secondary surgery was carried forward to the later time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Kyphoplasty | Vertebroplasty
Number analyzed (Participants) | 191 | 190
units on a scale
  Back pain at baseline (n=191, 190) | 7.8 (1.8) | 7.7 (1.8)
  Back pain at 7days (n=184, 180) | 4.2 (2.8) | 4.0 (2.5)
  Back pain at 30 days (n=169, 173) | 3.6 (2.9) | 3.5 (2.7)
  Back pain at 3 months (n=158, 156) | 3.3 (3.0) | 3.2 (2.8)
  Back pain at 12 months (n=142, 133) | 3.2 (3.0) | 3.5 (2.9)
  Back pain at 24 months (n=112, 108) | 3.7 (3.2) | 3.8 (3.0)
Statistical Analysis 1: Comparison: Kyphoplasty vs Vertebroplasty; Statistical analysis at 7 days; Test type: Superiority or Other; p = 0.430, ANCOVA — P-value was obtained from ANCOVA with baseline value as covariate
Statistical Analysis 2: Comparison: Kyphoplasty vs Vertebroplasty; Statistical analysis at 30 days; Test type: Superiority or Other; p = 0.655, ANCOVA — P-value was obtained from ANCOVA with baseline value as covariate
Statistical Analysis 3: Comparison: Kyphoplasty vs Vertebroplasty; Statistical analysis at 3 months; Test type: Superiority or Other; p = 0.756, ANCOVA — P-value was obtained from ANCOVA with baseline value as covariate
Statistical Analysis 4: Comparison: Kyphoplasty vs Vertebroplasty; Statistical analysis at 12 months; Test type: Superiority or Other; p = 0.503, ANCOVA — P-value was obtained from ANCOVA with baseline value as covariate
Statistical Analysis 5: Comparison: Kyphoplasty vs Vertebroplasty; Statistical analysis at 24 months; Test type: Superiority or Other; p = 0.837, ANCOVA — P-value was obtained from ANCOVA with baseline value as covariate

3. Secondary Outcome: Back Function-Oswestry Disability Index
Description: The Oswestry Disability Index (ODI) Questionnaire was used to assess patient back function. The ODI score ranges from 0-100. The best score is 0 (no disability) and worst is 100 (maximum disability).
Time Frame: 30 days, 3 months, 12 months, 24 months post-operation
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Kyphoplasty | Vertebroplasty
Number analyzed (Participants) | 191 | 190
units on a scale
  ODI at baseline (n=191, 189) | 59.0 (17.5) | 57.8 (16.0)
  ODI at 30 days (n=164, 156) | 36.2 (19.8) | 34.6 (17.6)
  ODI at 3 months (n=153, 141) | 30.4 (18.6) | 30.8 (18.0)
  ODI at 12 months (n=138, 119) | 29.2 (18.1) | 28.2 (17.8)
  ODI at 24 months (n=108, 93) | 32.1 (19.4) | 30.8 (17.8)
Statistical Analysis 1: Comparison: Kyphoplasty vs Vertebroplasty; Statistical analysis at 30 days; Test type: Superiority or Other; p = 0.785, ANCOVA — P-value was obtained from ANCOVA with baseline value as covariate
Statistical Analysis 2: Comparison: Kyphoplasty vs Vertebroplasty; Statistical analysis at 3 months; Test type: Superiority or Other; p = 0.393, ANCOVA — P-value was obtained from ANCOVA with baseline value as covariate
Statistical Analysis 3: Comparison: Kyphoplasty vs Vertebroplasty; Statistical analysis at 12 months; Test type: Superiority or Other; p = 0.875, ANCOVA — P-value was obtained from ANCOVA with baseline value as covariate
Statistical Analysis 4: Comparison: Kyphoplasty vs Vertebroplasty; Statistical analysis at 24 months; Test type: Superiority or Other; p = 0.833, ANCOVA — P-value was obtained from ANCOVA with baseline value as covariate

4. Secondary Outcome: Quality of Life by SF-36
Description: The Medical Outcomes Study 36-Item Short Form Health Survey (SF-36) was used to assess general health status. The SF-36 results are summarized into two components, a physical component summary (PCS) and a mental component summary (MCS). The score for PCS and MCS is between 0 and 100, with higher scores denoting better quality of life.
Time Frame: 30 days, 3 months, 12 months, 24 months post-operation
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Kyphoplasty | Vertebroplasty
Number analyzed (Participants) | 191 | 190
units on a scale
  SF-36 PCS at baseline (n=189, 190) | 27.92 (7.46) | 27.78 (8.20)
  SF-36 PCS at 30 days (n=162, 155) | 33.09 (10.13) | 34.51 (9.69)
  SF-36 PCS at 3 months (n=153, 138) | 36.06 (11.32) | 36.27 (10.66)
  SF-36 PCS at 12 months (n=138, 118) | 36.07 (11.33) | 37.39 (11.09)
  SF-36 PCS at 24 months (n=108, 92) | 34.94 (11.81) | 35.10 (9.98)
  SF-36 MCS at baseline (n=189, 190) | 40.87 (13.37) | 43.38 (12.73)
  SF-36 MCS at 30 days (n=162, 155) | 46.56 (12.83) | 47.43 (12.23)
  SF-36 MCS at 3 months (n=153, 138) | 49.86 (11.62) | 49.85 (11.16)
  SF-36 MCS at 12 months (n=138, 118) | 50.84 (11.75) | 49.99 (11.14)
  SF-36 MCS at 24 months (n=108, 92) | 48.84 (13.35) | 48.66 (12.24)
Statistical Analysis 1: Comparison: Kyphoplasty vs Vertebroplasty; Statistical analysis of SF-36 PCS result at 30 days; Test type: Superiority or Other; p = 0.180, ANCOVA — P-value was obtained from ANCOVA with baseline value as covariate
Statistical Analysis 2: Comparison: Kyphoplasty vs Vertebroplasty; Statistical analysis of SF-36 PCS result at 3 months; Test type: Superiority or Other; p = 0.822, ANCOVA — P-value was obtained from ANCOVA with baseline value as covariate
Statistical Analysis 3: Comparison: Kyphoplasty vs Vertebroplasty; Statistical analysis of SF-36 PCS result at 12 months; Test type: Superiority or Other; p = 0.291, ANCOVA — P-value was obtained from ANCOVA with baseline value as covariate
Statistical Analysis 4: Comparison: Kyphoplasty vs Vertebroplasty; Statistical analysis of SF-36 PCS result at 24 months; Test type: Superiority or Other; p = 0.996, ANCOVA — P-value was obtained from ANCOVA with baseline value as covariate
Statistical Analysis 5: Comparison: Kyphoplasty vs Vertebroplasty; Statistical analysis of SF-36 MCS result at 30 days; Test type: Superiority or Other; p = 0.983, ANCOVA — P-value was obtained from ANCOVA with baseline value as covariate
Statistical Analysis 6: Comparison: Kyphoplasty vs Vertebroplasty; Statistical analysis of SF-36 MCS result at 3 months; Test type: Superiority or Other; p = 0.576, ANCOVA — P-value was obtained from ANCOVA with baseline value as covariate
Statistical Analysis 7: Comparison: Kyphoplasty vs Vertebroplasty; Statistical analysis of SF-36 MCS result at 12 months; Test type: Superiority or Other; p = 0.393, ANCOVA — P-value was obtained from ANCOVA with baseline value as covariate
Statistical Analysis 8: Comparison: Kyphoplasty vs Vertebroplasty; Statistical analysis of SF-36 MCS result at 24 months; Test type: Superiority or Other; p = 0.722, ANCOVA — P-value was obtained from ANCOVA with baseline value as covariate

5. Secondary Outcome: Quality of Life -- EQ5D Index
Description: EQ-5D index scores range from 0 to 1.0 on a scale where 0 = death and 1.0 = perfect health.
Time Frame: 30 days, 3 months, 12 months, 24 months post-operation
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Kyphoplasty | Vertebroplasty
Number analyzed (Participants) | 191 | 190
units on a scale
  EQ5D index at baseline (n=189,189) | 0.44 (0.26) | 0.42 (0.24)
  EQ5D index at 30 days (n=164, 156) | 0.70 (0.19) | 0.71 (0.19)
  EQ5D index at 3 months (n=152, 140) | 0.75 (0.18) | 0.75 (0.17)
  EQ5D index at 12 months (n=137, 119) | 0.76 (0.18) | 0.77 (0.16)
  EQ5D index at 24 months (n=108, 94) | 0.72 (0.22) | 0.74 (0.19)
Statistical Analysis 1: Comparison: Kyphoplasty vs Vertebroplasty; Statistical analysis at 30 days; Test type: Superiority or Other; p = 0.318, ANCOVA — P-value was obtained from ANCOVA with baseline value as covariate
Statistical Analysis 2: Comparison: Kyphoplasty vs Vertebroplasty; Statistical analysis at 3 months; Test type: Superiority or Other; p = 0.523, ANCOVA — P-value was obtained from ANCOVA with baseline value as covariate
Statistical Analysis 3: Comparison: Kyphoplasty vs Vertebroplasty; Statistical analysis at 12 months; Test type: Superiority or Other; p = 0.634, ANCOVA — P-value was obtained from ANCOVA with baseline value as covariate
Statistical Analysis 4: Comparison: Kyphoplasty vs Vertebroplasty; Statistical analysis at 24 months; Test type: Superiority or Other; p = 0.457, ANCOVA — P-value was obtained from ANCOVA with baseline value as covariate

6. Secondary Outcome: Rate of Serious Adverse Events at 30 Days
Description: Rate of serious adverse events is presented as the percentage of the participants who reported serious adverse events within 30 days after initial treatment. For this study, serious adverse events (SAEs) included death, serious deterioration in health, life threatening injury/illness, hospitalization or prolonged hospitalization, or resulted in medical or surgical intervention.
Time Frame: 30 days post-operation
Population: Intent to treat population comprised of all subjects randomized and had initial treatment carried out.
Measure: Number; unit: percentage of participants
Arm/Group | Kyphoplasty | Vertebroplasty
Number analyzed (Participants) | 191 | 190
percentage of participants | 26.2 | 27.4
Statistical Analysis 1: Comparison: Kyphoplasty vs Vertebroplasty; Test type: Superiority or Other; p = 0.818, Fisher Exact

7. Primary Outcome: Percent of Subjects With One or More Subsequent Radiographic Fractures 24 Months
Time Frame: 24 months
Population: Intent to treat population comprised of all subjects randomized and had initial treatment carried out. The n for each group with available data at 24-months is indicated.
Measure: Number; unit: percentage of participants
Arm/Group | Kyphoplasty | Vertebroplasty
Number analyzed (Participants) | 110 | 111
percentage of participants
  No subsequence VCF | 50.9 | 42.3
  One or more subsequence VCFs | 49.1 | 57.7
Statistical Analysis 1: Comparison: Kyphoplasty vs Vertebroplasty; Test type: Superiority or Other; p = 0.226, Fisher Exact

8. Secondary Outcome: Rate of Procedure/Device Related or Possibly Related Serious Adverse Events at 30 Days
Description: Rate of Procedure/Device related or possibly related serious adverse events is presented as the percentage of the participants who reported Procedure/Device related or possibly related serious adverse events within 30 days after initial treatment.
Time Frame: 30 days post-operation
Population: Intent to treat population comprised of all subjects randomized and had initial treatment carried out.
Measure: Number; unit: percentage of participants
Arm/Group | Kyphoplasty | Vertebroplasty
Number analyzed (Participants) | 191 | 190
percentage of participants | 4.2 | 4.2
Statistical Analysis 1: Comparison: Kyphoplasty vs Vertebroplasty; Test type: Superiority or Other; p = 1.0, Fisher Exact

9. Secondary Outcome: Change in Anterior Vertebral Body Height
Time Frame: Pre-op, Pre-discharge, 3 months, 12 months, 24 months post-operation
Population: Intent to treat population comprised of all subjects randomized and had initial treatment carried out. The n for each group with available data (vertebrae) at each time point are indicated. The number of participants analyzed in 'Change in Anterior Vertebral Body Height' represents number of subjects with radiographic data available for analysis.
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: treated vertebrae
Arm/Group | Kyphoplasty | Vertebroplasty
Number analyzed (Participants) | 183 | 182
Number analyzed (treated vertebrae) | 232 | 224
mm
  Estimated Pre-Fracture (EP) height (n=231, 222) | 24.32 (3.93) | 24.49 (4.09)
  Vertebral body height at Pre-op (n=224, 212) | 15.91 (5.79) | 15.15 (6.04)
  Height Loss from EP/Absolute Height Loss (AHL) | -8.43 (4.47) | -9.22 (5.15)
  Change from pre-op to pre-discharge (n=217, 200) | 2.51 (3.19) | 2.40 (3.03)
  Change from pre-op to 3 months (n=176, 157) | 1.26 (2.99) | 1.23 (3.13)
  Change from pre-op to 12 months (n=158, 128) | 1.33 (3.12) | 1.05 (2.96)
  Change from pre-op to 24 months (n=101, 93) | 1.00 (3.08) | 0.75 (3.05)
Statistical Analysis 1: Comparison: Kyphoplasty vs Vertebroplasty; Statistical analysis at pre-discharge; Test type: Superiority or Other; p = 0.112, ANCOVA — P-value was obtained from ANCOVA with Absolute Height Loss (AHL) as covariate
Statistical Analysis 2: Comparison: Kyphoplasty vs Vertebroplasty; Statistical analysis at 3 months; Test type: Superiority or Other; p = 0.364, ANCOVA — P-value was obtained from ANCOVA with Absolute Height Loss (AHL) as covariate
Statistical Analysis 3: Comparison: Kyphoplasty vs Vertebroplasty; Statistical analysis at 12 months; Test type: Superiority or Other; p = 0.185, ANCOVA — P-value was obtained from ANCOVA with Absolute Height Loss (AHL) as covariate
Statistical Analysis 4: Comparison: Kyphoplasty vs Vertebroplasty; Statistical analysis at 24 months; Test type: Superiority or Other; p = 0.100, ANCOVA — P-value was obtained from ANCOVA with Absolute Height Loss (AHL) as covariate

10. Secondary Outcome: Change in Middle Vertebral Body Height
Time Frame: Pre-op, Pre-discharge, 3 months, 12 months, 24 months post-operation
Population: Intent to treat population comprised of all subjects randomized and had initial treatment carried out. The n for each group with available data (vertebrae) at each time point are indicated. The number of participants analyzed in 'Change in Middle Vertebral Body Height' represents number of subjects with radiographic data available for analysis.
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: treated vertebrae
Arm/Group | Kyphoplasty | Vertebroplasty
Number analyzed (Participants) | 183 | 182
Number analyzed (treated vertebrae) | 232 | 224
mm
  Estimated Pre-Fracture Height (EP) (n=231, 222) | 23.45 (3.46) | 23.68 (3.58)
  Vertebral body height at pre-op (n=225, 211) | 16.08 (5.08) | 15.92 (5.12)
  Height loss from EP/ Absolute Height Loss (AHL) | -7.42 (4.06) | -7.60 (4.09)
  change from pre-op at pre-discharge (n=219, 200) | 2.33 (2.72) | 1.84 (2.38)
  Change from pre-op at 3 months (n=177, 159) | 1.34 (2.59) | 1.18 (2.55)
  Change from pre-op at 12 months (n=161, 128) | 1.31 (2.80) | 0.92 (2.51)
  Change from pre-op at 24 months (n=104, 92) | 0.98 (2.58) | 0.67 (2.78)
Statistical Analysis 1: Comparison: Kyphoplasty vs Vertebroplasty; Statistical analysis at pre-discharge; Test type: Superiority or Other; p = 0.005, ANCOVA — P-value was obtained from ANCOVA with Absolute Height Loss (AHL) as covariate
Statistical Analysis 2: Comparison: Kyphoplasty vs Vertebroplasty; Statistical analysis at 3 months; Test type: Superiority or Other; p = 0.382, ANCOVA — P-value was obtained from ANCOVA with Absolute Height Loss (AHL) as covariate
Statistical Analysis 3: Comparison: Kyphoplasty vs Vertebroplasty; Statistical analysis at 12 months; Test type: Superiority or Other; p = 0.196, ANCOVA — P-value was obtained from ANCOVA with Absolute Height Loss (AHL) as covariate
Statistical Analysis 4: Comparison: Kyphoplasty vs Vertebroplasty; Statistical analysis at 24 months; Test type: Superiority or Other; p = 0.281, ANCOVA — P-value was obtained from ANCOVA with Absolute Height Loss (AHL) as covariate

11. Secondary Outcome: Change in Posterior Vertebral Body Height
Time Frame: Pre-op, Pre-discharge, 3 months, 12 months, 24 months post-operation
Population: Intent to treat population comprised of all subjects randomized and had initial treatment carried out. The n for each group with available data (vertebrae) at each time point are indicated. The number of participants analyzed in 'Change in Posterior Vertebral Body Height' represents number of subjects with radiographic data available for analysis.
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: treated vertebrae
Arm/Group | Kyphoplasty | Vertebroplasty
Number analyzed (Participants) | 183 | 182
Number analyzed (treated vertebrae) | 232 | 224
mm
  Estimated Pre-Fracture Height (n=231, 222) | 25.89 (3.45) | 26.10 (3.67)
  Vertebral body height at pre-op (n=225, 210) | 23.41 (4.11) | 23.47 (4.36)
  Height Loss from EP/Absolute Height Loss (AHL) | -2.52 (2.47) | -2.49 (2.46)
  Change from pre-op to pre-discharge (n=220, 199) | 0.82 (1.74) | 0.49 (1.50)
  Change from pre-op to 3 months (n=179, 160) | 0.10 (1.64) | 0.06 (1.63)
  Change from pre-op to 12 months (n=161, 129) | -0.03 (1.79) | -0.00 (1.78)
  Change from pre-op to 24 months (n=104, 93) | -0.21 (1.55) | -0.30 (1.79)
Statistical Analysis 1: Comparison: Kyphoplasty vs Vertebroplasty; Statistical analysis at pre-discharge; Test type: Superiority or Other; p = 0.033, ANCOVA — P-value was obtained from ANCOVA with Absolute Height Loss (AHL) as covariate
Statistical Analysis 2: Comparison: Kyphoplasty vs Vertebroplasty; Statistical analysis at 3 months; Test type: Superiority or Other; p = 0.981, ANCOVA — P-value was obtained from ANCOVA with Absolute Height Loss (AHL) as covariate
Statistical Analysis 3: Comparison: Kyphoplasty vs Vertebroplasty; Statistical analysis at 12 months; Test type: Superiority or Other; p = 0.631, ANCOVA — P-value was obtained from ANCOVA with Absolute Height Loss (AHL) as covariate
Statistical Analysis 4: Comparison: Kyphoplasty vs Vertebroplasty; Statistical analysis at 24 months; Test type: Superiority or Other; p = 0.790, ANCOVA — P-value was obtained from ANCOVA with Absolute Height Loss (AHL) as covariate

12. Secondary Outcome: Change in Vertebral Body Kyphosis Angle
Description: The vertebral kyphosis angle was defined as the angle formed by lines drawn parallel to the superior and inferior endplates of the treated fractured vertebral body.
Time Frame: Pre-op, Pre-discharge, 3 months, 12 months, 24 months post-operation
Population: Intent to treat population comprised of all subjects randomized and had initial treatment carried out. The n for each group with available data (vertebrae) at each time point are indicated. The number of participants analyzed in 'Change in Vertebral Body Kyphosis Angle' represents number of subjects with radiographic data available for analysis.
Measure: Mean (Standard Deviation); unit: degree
Units Other Than Participants: treated vertebrae
Arm/Group | Kyphoplasty | Vertebroplasty
Number analyzed (Participants) | 183 | 182
Number analyzed (treated vertebrae) | 232 | 224
degree
  Kyphosis angle at pre-op (n=219, 210) | -14.17 (8.29) | -15.68 (8.12)
  Change from pre-op to pre-discharge (n=213, 195) | 3.10 (5.22) | 3.41 (5.67)
  Change from pre-op to 3 months (n=168, 155) | 1.78 (5.25) | 2.28 (5.72)
  Change from pre-op to 12 months (n=154, 127) | 1.97 (5.38) | 1.51 (5.30)
  Change from pre-op to 24 months (n=99, 92) | 2.09 (5.95) | 1.43 (5.01)
Statistical Analysis 1: Comparison: Kyphoplasty vs Vertebroplasty; Statistical analysis at pre-discharge; Test type: Superiority or Other; p = 0.663, ANCOVA — P-value was obtained from ANCOVA with baseline value as covariate
Statistical Analysis 2: Comparison: Kyphoplasty vs Vertebroplasty; Statistical analysis at 3 months; Test type: Superiority or Other; p = 0.933, ANCOVA — P-value was obtained from ANCOVA with baseline value as covariate
Statistical Analysis 3: Comparison: Kyphoplasty vs Vertebroplasty; Statistical analysis at 12 months; Test type: Superiority or Other; p = 0.089, ANCOVA — P-value was obtained from ANCOVA with baseline value as covariate
Statistical Analysis 4: Comparison: Kyphoplasty vs Vertebroplasty; Statistical analysis at 24 months; Test type: Superiority or Other; p = 0.036, ANCOVA — P-value was obtained from ANCOVA with baseline value as covariate

13. Secondary Outcome: Change in Vertebral Body Local Cobb Angle (LCA)
Description: The vertebral body local Cobb angle is a measurement of the 3-level functional unit consisting of the treated fractured vertebral body and the nearest adjacent vertebrae and is defined as the angle formed by lines drawn parallel to the superior endplate of the cranial adjacent vertebral body and the inferior endplate of the adjacent caudal vertebral body.
Time Frame: Pre-op, Pre-discharge, 3 months, 12 months, 24 months post-operation
Population: Intent to treat population comprised of all subjects randomized and had initial treatment carried out. The n for each group with available data (vertebrae) at each time point are indicated. The number of participants analyzed in 'Change in Vertebral Body Local Cobb Angle' represents number of subjects with radiographic data available for analysis.
Measure: Mean (Standard Deviation); unit: degree
Units Other Than Participants: treated vertebrae
Arm/Group | Kyphoplasty | Vertebroplasty
Number analyzed (Participants) | 183 | 182
Number analyzed (treated vertebrae) | 232 | 224
degree
  Vertebral body LCA at pre-op (n=213, 203) | -14.00 (19.71) | -15.48 (18.67)
  Change from pre-op to pre-discharge (n=203, 186) | 2.37 (5.84) | 2.84 (4.33)
  Change from pre-op to 3 months (n=166, 146) | -0.22 (5.46) | -0.43 (6.67)
  Change from pre-op to 12 months (n=151, 118) | 0.38 (10.15) | 0.03 (8.15)
  Change from pre-op to 24 months (n=98, 85) | -1.15 (8.43) | -0.57 (6.35)
Statistical Analysis 1: Comparison: Kyphoplasty vs Vertebroplasty; Statistical analysis at pre-discharge; Test type: Superiority or Other; p = 0.472, ANCOVA — P-value was obtained from ANCOVA with baseline value as covariate
Statistical Analysis 2: Comparison: Kyphoplasty vs Vertebroplasty; Statistical analysis at 3 months; Test type: Superiority or Other; p = 0.745, ANCOVA — P-value was obtained from ANCOVA with baseline value as covariate
Statistical Analysis 3: Comparison: Kyphoplasty vs Vertebroplasty; Statistical analysis at 12 months; Test type: Superiority or Other; p = 0.565, ANCOVA — P-value was obtained from ANCOVA with baseline value as covariate
Statistical Analysis 4: Comparison: Kyphoplasty vs Vertebroplasty; Statistical analysis at 24 months; Test type: Superiority or Other; p = 0.687, ANCOVA — P-value was obtained from ANCOVA with baseline value as covariate

14. Secondary Outcome: Change in Global Sagittal Balance.
Description: Change in global sagittal balance as measured by sagittal vertical axis.
Time Frame: Pre-op, Pre-discharge, 3 months, 12 months, 24 months post-operation
Population: Due to the early termination of the study and having few sites able to image using 3-foot lateral films, sponsor will not carry out the analysis of global sagittal balance in the clinic report.
Arm/Group | Kyphoplasty | Vertebroplasty
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: VCF-related Health Care Utilization
Description: Health care utilization assessments conducted by monthly phone call to participating patients.
Time Frame: Monthly for 24 months post-op
Population: Due to the early termination of the study, sponsor will not carry out the analysis of secondary healthcare utilization endpoints.
Arm/Group | Kyphoplasty | Vertebroplasty
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 24 months
Description: For this study, serious adverse events (SAEs) included death, serious deterioration in health, life threatening injury/illness, hospitalization or prolonged hospitalization, or resulted in medical or surgical intervention.
Arm/Group | Kyphoplasty | Vertebroplasty
Serious Adverse Events (participants affected / at risk) | 125/191 | 125/190
Other Adverse Events (participants affected / at risk) | 55/191 | 69/190
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Kyphoplasty (N=191) | Vertebroplasty (N=190)
Anaemia (Blood and lymphatic system disorders) | 6 (7) | 4 (4)
Coagulopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Heparin-induced thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Polycythaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 2 (2) | 3 (3)
Aortic valve stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 6 (7) | 5 (5)
Cardiac arrest (Cardiac disorders) | 1 (2) | 3 (4)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 6 (6) | 10 (18)
Cardio-respiratory arrest (Cardiac disorders) | 2 (2) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Chest pain (Cardiac disorders) | 1 (1) | 1 (1)
Coronary artery disease (Cardiac disorders) | 2 (2) | 1 (1)
Coronary artery occlusion (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Heart valve incompetence (Cardiac disorders) | 1 (1) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 1 (1) | 1 (1)
Myocardial infarction (Cardiac disorders) | 4 (5) | 3 (3)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 2 (2)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Cerumen impaction (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Deafness neurosensory (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Hearing impaired (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 3 (3) | 3 (4)
Conjunctival haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Diplopia (Eye disorders) | 0 (0) | 1 (1)
Sjogren's syndrome (Eye disorders) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
abdominal pain (Gastrointestinal disorders) | 1 (1) | 6 (6)
abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 2 (3) | 2 (2)
Colitis ulcerative (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 4 (5) | 6 (6)
Crohn's disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric polyps (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 5 (5)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus paralytic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Impaired gastric emptying (Gastrointestinal disorders) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 2 (2) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 5 (6)
Oesophageal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatic cyst (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 2 (2) | 1 (1)
Rectal prolapse (Gastrointestinal disorders) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3) | 5 (6)
Peptic ulcer (Gastrointestinal disorders) | 0 (0) | 2 (2)
Proctitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Adverse drug reaction (General disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 1 (2) | 1 (1)
Chest pain (General disorders) | 0 (0) | 4 (4)
Death (General disorders) | 2 (2) | 3 (3)
Generalised oedema (General disorders) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 3 (3) | 0 (0)
Oedema peripheral (General disorders) | 2 (2) | 4 (5)
Pain (General disorders) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 2 (3)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 1 (1)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis chronic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 2 (2) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1) | 1 (1)
Abscess (Infections and infestations) | 0 (0) | 1 (1)
Abscess oral (Infections and infestations) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 10 (11) | 7 (11)
Cellulitis (Infections and infestations) | 3 (4) | 3 (3)
Clostridial infection (Infections and infestations) | 1 (1) | 2 (2)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 1 (1)
Corynebacterium infection (Infections and infestations) | 1 (1) | 0 (0)
Encephalitis viral (Infections and infestations) | 1 (1) | 0 (0)
Endocarditis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 3 (3) | 0 (0)
Gastroenteritis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 2 (3) | 1 (1)
Herpes zoster (Infections and infestations) | 2 (2) | 0 (0)
Hordeolum (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 2 (2)
Localised infection (Infections and infestations) | 2 (2) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Onychomycosis (Infections and infestations) | 0 (0) | 2 (2)
Otitis media (Infections and infestations) | 1 (1) | 0 (0)
Otitis media chronic (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 14 (16) | 12 (18)
Pneumonia pneumococcal (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Sepsis syndrome (Infections and infestations) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 1 (1) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 2 (2)
Skin infection (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal abscess (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 0 (0) | 2 (2)
Streptococcal infection (Infections and infestations) | 0 (0) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 6 (7) | 6 (6)
Urinary tract infection (Infections and infestations) | 10 (16) | 18 (24)
Urinary tract infection enterococcal (Infections and infestations) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
Accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Acetabulum fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Arthropod sting (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Back injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Bone fissure (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Burns second degree (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Catheter site haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cement embolism (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 2 (2) | 4 (4)
Dural tear (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 30 (44) | 32 (39)
Femur fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 2 (3) | 2 (2)
Fractured sacrum (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 5 (5) | 5 (5)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Joint sprain (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Low limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Mental status changes postoperative (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 4 (4) | 3 (3)
Peripheral nerve injury (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural hypotension (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Procedural nausea (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 7 (7) | 7 (8)
Procedural vomiting (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pubis fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 7 (7) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 3 (3) | 2 (3)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Spinal fracture (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Tibia fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Traumatic brain injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Wound haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 4 (4) | 0 (0)
Aspiration tracheal (Investigations) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0)
White blood cell count increased (Investigations) | 1 (1) | 0 (0)
Abnormal loss weight (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Adrenal insufficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 5 (6) | 2 (2)
Diabetic complication (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Fluid retention (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Gout (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypovolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Shock hypoglycaemic (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 15 (22) | 7 (8)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Arthropathy (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 42 (63) | 42 (69)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bunion (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Congenital jaw malformation (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Contusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Facet joint syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Gout (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Groin pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Iliotibial band syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (3)
Lumbar vertebral fracture (Musculoskeletal and connective tissue disorders) | 9 (13) | 13 (18)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (4)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 5 (7) | 5 (6)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 5 (5)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (6)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (4) | 8 (9)
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Restless legs syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Sacroiliitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Sinus tarsi syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Spinal fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Thoracic vertebral fracture (Musculoskeletal and connective tissue disorders) | 19 (24) | 19 (29)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Anal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Endometrial cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Monoclonal gammopathy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Paraproteinaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Polyp (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Small intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Amnesia (Nervous system disorders) | 0 (0) | 1 (1)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 5 (5) | 2 (2)
Convulsion (Nervous system disorders) | 1 (1) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 5 (7)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (3) | 5 (6)
Intracranial aneurysm (Nervous system disorders) | 0 (0) | 1 (1)
Lethargy (Nervous system disorders) | 2 (2) | 1 (1)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Lumbar radiculopathy (Nervous system disorders) | 0 (0) | 1 (2)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Parkinson's disease (Nervous system disorders) | 0 (0) | 1 (1)
Piriformis syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Radicular pain (Nervous system disorders) | 2 (2) | 2 (2)
Sciatica (Nervous system disorders) | 1 (1) | 2 (2)
Spinal cord compression (Nervous system disorders) | 1 (1) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 3 (3)
Toxic neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1)
Abnormal behaviour (Psychiatric disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 2 (3) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1)
Dementia (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 4 (5) | 1 (1)
Hallucination (Psychiatric disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (2) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 3 (5)
Hypertonic bladder (Renal and urinary disorders) | 0 (0) | 1 (1)
Ketonuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Polyuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 4 (4) | 1 (1)
Renal failure chronic (Renal and urinary disorders) | 2 (3) | 1 (1)
Renal pain (Renal and urinary disorders) | 1 (1) | 0 (0)
Stress urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
Ureteric stenosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Urge incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 3 (3) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 1 (1) | 2 (3)
Uterine prolapse (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (5)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 5 (9) | 8 (11)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (6)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Oropharyngeal blistering (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 2 (2)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sleep apnea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dyshidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pemphigoid (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 2 (3) | 1 (1)
Adenotonsillectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Cataract operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Coronary angioplasty (Surgical and medical procedures) | 1 (1) | 0 (0)
Knee arthroplasty (Surgical and medical procedures) | 0 (0) | 1 (1)
Small intestinal resection (Surgical and medical procedures) | 0 (0) | 1 (1)
Spinal laminectomy (Surgical and medical procedures) | 0 (0) | 1 (2)
Aortic aneurysm (Vascular disorders) | 2 (2) | 0 (0)
Aortic dissection (Vascular disorders) | 1 (1) | 0 (0)
Carotid artery stenosis (Vascular disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 3 (3) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 2 (3) | 0 (0)
Intermittent claudication (Vascular disorders) | 1 (1) | 1 (1)
Lymphoedema (Vascular disorders) | 1 (1) | 1 (1)
Migraine (Vascular disorders) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 2 (2)
Peripheral vascular disorder (Vascular disorders) | 1 (1) | 1 (1)
Venous insufficiency (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Kyphoplasty (N=191) | Vertebroplasty (N=190)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Bone marrow oedema (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Mitral valve incompetence (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Eustachian tube dysfunction (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Inner ear disorder (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Goitre (Endocrine disorders) | 1 (1) | 1 (1)
Vitreous detachment (Eye disorders) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Frequent bowel movements (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Retching (Gastrointestinal disorders) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Asthenia (General disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 1 (1)
Injection site haematoma (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 3 (3)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2)
Viral infection (Infections and infestations) | 0 (0) | 1 (1)
Acetabulum fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Back injury (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Back pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 2 (3) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 23 (28) | 20 (24)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ilium fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Implant site extravasation (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Joint sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post-traumatic pain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 5 (5) | 2 (2)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 4 (4)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Skeletal injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Soft tissue injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Immunoglobulins increased (Investigations) | 1 (1) | 0 (0)
Abnormal loss of weight (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Adrenal insufficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 5 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 9 (10) | 19 (20)
Coccydynia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Facet joint syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Lumbar vertebral fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Muscle strain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Spinal fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Thoracic vertebral fracture (Musculoskeletal and connective tissue disorders) | 3 (4) | 3 (3)
Vaginal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 2 (2)
Grand mal convulsion (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 2 (2) | 3 (3)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 1 (1)
Nystagmus (Nervous system disorders) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Polyneuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 1 (1)
Vocal cord paralysis (Nervous system disorders) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (2) | 0 (0)
Ovarian mass (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The original study design required n=1,234 randomized patients; however, the study was stopped early with only n=404 enrolled patients, due to low enrollment, difficulty in willingness to randomize patients and a high proportion of early terminations

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less